CLINICAL TRIAL: NCT01578824
Title: Assessment Of Vitamin D Role In The Pathogenesis Of Asthma In Vitamin D Resistent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Vit D and asthma in VDRR CTIL
Record Dates: First submitted 2011-11-09; First posted 2012-04-17 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Asthma; Vitamin D Resistant Rickets
Keywords: Rickets; Vitamin D; airway hyperreactivity; Exhaled breath condensate
MeSH Terms: conditions — Asthma; Familial Hypophosphatemic Rickets; Rickets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Control (Active Comparator)
  Interventions: Other: Methacholine Challenge Test
- Vitamin D resistant Rickets (Active Comparator): Vitamin D resistant Rickets patients
  Interventions: Other: Methacholine Challenge Test

INTERVENTIONS:
Other: Methacholine Challenge Test — Evaluation of airway hyperreactivity as assessed by doubling dose of methacholine with determination of PC20
  Other Names: Airway Hyperresponsiveness test

SUMMARY:
Research Title: Evaluation of airway reactivity, allergy and inflammatory mediators in exhaled breath condensate in vitamin D resistant rickets.

Aim: To assess the effect of absence of vitamin D receptors on airway reactivity, allergy and inflammatory mediators in exhaled breath condensate in a prospective study evaluating patients with vitamin D resistant rickets and in healthy controls.

Sample size: 40 participants in the two groups. Primary end point: Airway reactivity as assessed by methacholine challenge test.

Secondary outcome parameters: All other parameters are the secondary end points.

DETAILED DESCRIPTION:
Research Title: Evaluation of airway reactivity, allergy and inflammatory mediators in exhaled breath condensate in vitamin D resistant rickets.

Introduction: Vitamin D seems to play a role in allergic and asthmatic reactions. Vitamin D resistant rickets patients lack vitamin D receptors and cannot absorb vitamin D.

Aim: To assess the effect of absence of vitamin D receptors on airway reactivity, allergy and inflammatory mediators in exhaled breath condensate.

Design: Prospective study evaluating these parameters in patients with vitamin D resistant rickets and in healthy controls.

Participant selection: The study group will consist of vitamin D resistant rickets patients followed and treated at the Pediatric Endocrinology Department at our hospital. The study group will be compared to an age- and sex-matched healthy control group that had a negative methacholine challenge test.

Sample size: 40 participants in the two groups. Intervention: Each subject will undergo evaluation including a respiratory questionnaire, pulmonary function tests, methacholine challenge test with determination of PC20, exhaled nitric oxide (eNO), and exhaled breath condensate (EBC). Venous blood will be analyzed for complete blood count + eosinophils, IGE levels, and Vitamin D levels. Prick skin test for inhaled allergens will be performed. All measurements will be evaluated in a single 3 hour visit, with no follow up study visits.

Primary end point: Airway reactivity as assessed by methacholine challenge test.

Secondary outcome parameters: All other parameters are the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D Resistent Rickets
* Age between 3 - 40 years

Exclusion Criteria:

* Any Chronic Lung Disease
* Febrile Illness in last 2 weeks
* Inhaled Corticosteroids over the past 2 weeks
* Bronchodilators over the past 24 hours
* Participation in any other clinical studies over the past 4 weeks

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Metacholine Challenge Test | participants will be followed for the duration of hospital visit, an average of 3 hours
  As assessed by methacholine challenge test with determination of PC20.

SECONDARY OUTCOMES:
IgE | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count
CBC | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count
Fractional Exhaled NO | participants will be followed for the duration of hospital visit, an average of 3 hours
  determination of exhaled NO in Exhaled breath
skin tests for inhaled allergens | participants will be followed for the duration of hospital visit, an average of 3 hours
Inhaled breath condensate | participants will be followed for the duration of hospital visit, an average of 3 hours
C reactive protein | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count
25 OH vitamin D3 | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam MC
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel, Israel